CLINICAL TRIAL: NCT06042010
Title: Efficacy of Oral Zinc Supplement as an Adjunctive Therapy for Erosive Oral Lichen Planus (a Randomized, Controlled Clinical Trial)
Brief Title: Oral Zinc Supplement as Adjunctive Therapy for Erosive Oral Lichen Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Oral medicine_0424-04\2022
Record Dates: First submitted 2023-09-12; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental)
  Interventions: Drug: Oral zinc supplement
- control group (Active Comparator)
  Interventions: Drug: triamcinolone acetonide Oral paste

INTERVENTIONS:
Drug: Oral zinc supplement — patients received oral Zinc picolinate 50mg for 6 weeks as single morning dose along with 0.1%
  Arms: Test group
Drug: triamcinolone acetonide Oral paste — patients will received 0.1%triamcinolone acetonide Oral paste twice daily alone for 6weeks.
  Arms: control group

SUMMARY:
Lichen Planus (LP) is a chronic mucocutaneous inflammatory disease and considered as T-cell mediated autoimmune disorder.

Zinc is a potent antioxidant micronutrient that contributes to the proper functioning of the antioxidant defense system. In addition, this mineral protects cells against inflammation by oxidative stress, because it acts in the stabilization of cell membrane. It also maintains macrophage and neutrophil functions, natural killer cell activity, and complement activity.

Matrix metalloproteinases (MMPs) are a family of zinc-containing endopeptidases and have the main function of proteolytic degradation of connective tissue matrix proteins. Zinc prevents (MMP-1) activation and inhibition of the T-cell accumulation in (OLP) through inhibiting of (MMP-9).

Aim of the study: To evaluate and compare the efficacy of adding oral zinc supplementation 50 mg to 0.1%Triamcinolone orabase (TA)versus 0.1%Triamcinolone orabase alone on the healing of erosive OLP.

ELIGIBILITY:
Inclusion Criteria:

* All patients involved in this clinical trial will have symptomatic OLP

Exclusion Criteria:

* Smokers or tobacco users will be excluded from this clinical trial.
* Pregnant and lactating females.
* Any patient that has history of cancer, kidney, liver or other autoimmune disease will be excluded from this study.
* Patients showing dysplastic changes in their confirmatory biopsy specimen will be also excluded.
* Any patients presenting with extra oral lichen planus lesions will be excluded.
* Suspicious lesions of both lichenoid contact reaction and lichenoid drug reaction lesions will be excluded.
* Vitamin administration intake within the last 3 months

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Change in oral lesions | Baseline, 6 weeks, 12 weeks
  Thongprasom scoring system will be used for the measurement of objective outcomes; score 5 was assigned to patients having white striae with erosive areas >1 cm2, score 4 assigned to patients with white striae and erosive areas <1 cm2, score 3 assigned to those having white striae and atrophic areas >1 cm2, score 2 assigned to those having white striae and atrophic areas <1 cm2, score 1 assigned to those having only white striae, and score 0 assigned to normal mucosa.
Change in MMP-9 level | Baseline, 6 weeks, 12 weeks
  Whole unstimulated saliva will be collected from all participants

SECONDARY OUTCOMES:
Change in pain | Baseline, 6 weeks, 12 weeks
  Patients will be asked to assign a numerical score representing the intensity of their symptoms on a scale from 0 to 10, with 0 being no symptoms and 10 being worst imaginable symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt